CLINICAL TRIAL: NCT01926106
Title: Nasal Intermittent Positive-Pressure Ventilation vs Nasal Continuous Positive Airway Pressure for Twin Infants With Respiratory Distress Syndrome
Brief Title: Nasal Intermittent Positive-Pressure Ventilation for Twin Infants With Respiratory Distress Syndrome
Acronym: twins
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Daping Hospital and the Research Institute of Surgery of the Third Military Medical University (Other)
Responsible Party: Principal Investigator, Chen Long,MD, Prof;MD, Daping Hospital and the Research Institute of Surgery of the Third Military Medical University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: twins
Record Dates: First submitted 2013-08-08; First posted 2013-08-20 (Estimated); Last update posted 2017-12-07 (Actual); Status verified 2013-08

CONDITIONS: Neonatal Respiratory Distress Syndrome
Keywords: Nasal Intermittent Positive-Pressure Ventilation; Nasal Continuous Positive Airway Pressure; twin; respiratory distress syndrome
MeSH Terms: conditions — Respiratory Distress Syndrome, Newborn; Respiratory Distress Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- nIPPV (Experimental): the infants in the arm were supported by Nasal Intermittent Positive-Pressure Ventilation(nIPPV)
  Interventions: Device: nIPPV
- nCPAP (Active Comparator): the infants in the arm were supported by Nasal Continuous Positive Airway Pressure(nCPAP)
  Interventions: Device: nCPAP

INTERVENTIONS:
Device: nIPPV — one of the twins was randomly allocated to nIPPV
  Other Names: nIPPV:Nasal Intermittent Positive Pressure Ventilation
  Arms: nIPPV
Device: nCPAP — another of the twins was allocated to nCPAP
  Other Names: nCPAP:Nasal Continuous Positive Airway Pressure
  Arms: nCPAP

SUMMARY:
In the present study, we hypothesized that primary mode nIPPV initiated shortly after birth would decrease the incidence of intubation or death in twin infants when compared to nCPAP.

DETAILED DESCRIPTION:
After inclusion of eligible twins infants,one of the twins was supported by nCPAP and another nIPPV.

ELIGIBILITY:
Inclusion Criteria:

* Twins
* Clinical diagnosis of mild-moderate respiratory distress syndrome
* requiring a fraction of inspired oxigen (FiO2 ) <0.40 to keep oxygen saturation of 90%-95%
* a chest X-ray suggestive of early stage hyaline membrane disease, (i.e. mild microgranulia and air bronchogram)

Exclusion Criteria:

* pneumothorax
* pneumomediastinum
* surgical diseases
* cardiac diseases
* intraventricular hemorrage
* major congenital defects

Ages: 30 Minutes to 6 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 286 (Actual)
Dates: Start 2012-07-01 (Actual); Primary Completion 2017-07-30 (Actual); Study Completion 2017-07-30 (Actual)

PRIMARY OUTCOMES:
incidence of intubation | 48h

SECONDARY OUTCOMES:
incidence of BPD | 1 month

OTHER OUTCOMES:
death | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Long Chen, MD, Principal Investigator — Department of Pediatrics, Daping Hospital, Research Institute of Surgery, Third Military Medical University,
Locations (1):
- Department of Pediatrics, Daping Hospital, Research Institute of Surgery, Third Military Medical University, Chongqing, Chongqing Municipality, China